CLINICAL TRIAL: NCT06110910
Title: Long-term Efficacy and Safety Evaluation of Growth Hormone in Children in China(CGLS)-an Open-label, Multicenter, Prospective and Retrospective Observational Study
Brief Title: Long-term Efficacy and Safety Evaluation of Growth Hormone in Children in China(CGLS)
Status: Recruiting | Type: Observational
Sponsor: Xiaoping Luo (Other)
Responsible Party: Sponsor-Investigator, Xiaoping Luo, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202410048
Record Dates: First submitted 2023-10-07; First posted 2023-11-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Childhood Short Stature
MeSH Terms: interventions — polyethylene glycol-recombinant human growth hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- prospective cohort: Polvethylene glycol recombinant human growth hormone injection (PEG-rhGH) and recombinanthuman growth hormone injection (rhGH) were used.
  Interventions: Drug: Polvethylene glycol recombinant human growth hormone injection (PEG-rhGH) or recombinanthuman growth hormone injection (rhGH)
- retrospective cohort: Polvethylene glycol recombinant human growth hormone injection (PEG-rhGH) and recombinanthuman growth hormone injection (rhGH) were used.
  Interventions: Drug: Polvethylene glycol recombinant human growth hormone injection (PEG-rhGH) or recombinanthuman growth hormone injection (rhGH)
- ambispective cohort: Polvethylene glycol recombinant human growth hormone injection (PEG-rhGH) and recombinanthuman growth hormone injection (rhGH) were used.
  Interventions: Drug: Polvethylene glycol recombinant human growth hormone injection (PEG-rhGH) or recombinanthuman growth hormone injection (rhGH)

INTERVENTIONS:
Drug: Polvethylene glycol recombinant human growth hormone injection (PEG-rhGH) or recombinanthuman growth hormone injection (rhGH) — Polvethylene glycol recombinant human growth hormone injection (PEG-rhGH) and recombinanthuman growth hormone injection (rhGH) were used.
  Other Names: PEG-rhGH or rhGH

SUMMARY:
Short stature is a relatively common pediatric condition, referring to individuals whose height is more than 2 (-2 SD) standard deviations below the average height of a similar age, gender, and ethnicity population in similar living conditions, or those below the third percentile (-1.88 SD). This study is an open-label, multicenter, prospective and retrospective, observational, cohort study aimed at assessing the long-term safety and efficacy of PEG-rhGH or rhGH treatment for Chinese children with short stature. The study is divided into retrospective cohorts, retrospective prospective cohorts, and prospective cohorts. It is expected to include approximately 10000 patients (including around 3000 in the retrospective cohorts and around 7000 in the retrospective prospective and prospective cohorts). The total duration is expected to be 16 years, including 2 years for study center initiation and patient recruitment and follow-up of patients in the retrospective prospective and prospective cohorts until near-adult height (NAH). The primary objective is to evaluate the long-term safety of PEG-rhGH or rhGH for the treatment of children with short stature (including GHD, ISS, SGA, TS, PWS, NS, SHOX gene deletion, and other etiologies); the secondary objective is to assess the effectiveness of PEG-rhGH or rhGH treatment for children with short stature (including GHD, ISS, SGA, TS, PWS, NS, SHOX gene deletion, and other etiologies).

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2 years and older with various causes of short stature.
2. Height below the 3rd percentile (-1.88 SD) compared to the height of normal, healthy children of the same age and gender.
3. Belonging to one of the following indications: GHD, ISS, SGA, TS, PWS, NS, SHOX gene deletion, or other causes of short stature.

Note: In this study, the inclusion criteria for the PWS cohort do not impose restrictions on height and age at the start of treatment.

Exclusion Criteria:

1. Patients with fully closed growth plates.
2. Patients with signs of potential tumor progression or those already diagnosed with tumors.
3. Allergic reactions to growth hormone or its adjuvants.
4. Patients who have received any growth hormone treatment other than the investigational drug in the six months prior to screening.
5. Any other circumstances deemed unsuitable for study inclusion by the investigator.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Childhood short stature includes various conditions such as Growth Hormone Deficiency (GHD), Idiopathic Short Stature (ISS), Small for Gestational Age (SGA), Turner Syndrome (TS), Prader-Willi Syndrome (PWS), Noonan Syndrome (NS), SHOX gene deletion, and other causes of short stature.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The AE (Adverse Event) and SAE (Serious Adverse Event) occurrence rates | From the time of signing the informed consent form to the near adult height(NAH), the overall assessment time was approximately 192 months.
  An adverse event refers to any unfavorable medical occurrence in a patient after receiving the investigational drug, which can manifest as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily be causally related to the investigational drug. SAE, on the other hand, stands for serious adverse events, which encompass events such as patient death, life-threatening situations, permanent or severe disabilities or functional loss, hospitalization or extended hospital stays, as well as congenital anomalies or birth defects, among other adverse medical occurrences, following the administration of the investigational drug.

CONTACTS AND LOCATIONS:
Overall Officials: xiaoping Luo, doctor, Principal Investigator — Tongji Hospital
Locations (1):
- TongjiHospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Wu W, Luo X. Long-Term Efficacy and Safety of Growth Hormone in Children Suffering from Short Stature in China (CGLS): An Open-Label, Multicenter, Prospective and Retrospective, Observational Study. Adv Ther. 2025 Jun;42(6):2957-2969. doi: 10.1007/s12325-025-03146-2. Epub 2025 Apr 8. PMID 40198521